CLINICAL TRIAL: NCT00379314
Title: A Randomized, Prospective, Multicenter Trial Comparing TVT With TVT-O Procedures in Treatment of Female Primary Urinary Stress Incontinence
Brief Title: Randomized, Multicenter Trial Comparing TVT With TVT-O for Treatment of Female Urinary Incontinence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42/E8/04
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-09

CONDITIONS: Urinary Stress Incontinence
Keywords: Incontinence; Urinary; Female; Surgery; Complications
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Procedure: TVT and TVT-O minimally invasive surgical procedures
Procedure: Surgery for female stress urinary incontinence

SUMMARY:
The Tensionfree Vaginal Tape (TVT) procedure is a minimally invasive surgical procedure for treatment of female urinary stress incontinence. The TVT procedure has a documented efficacy and safety but is still associated with the risk of intra- and post-operative complications. A modification of the TVT procedure called TVT-O (Tensionfree Vaginal Tape Obturator), which utilises the obturator foramen for passage of the tape, is thought to lower the risk of complications. The trial compares the TVT procedure with the TVT-O procedure in a randomized fashion in order to detect differences in the rate of complications and in cure rate.

ELIGIBILITY:
Inclusion Criteria:

* history of stress incontinence
* indications for surgical treatment
* positive cough stress test
* urgency score < 7

Exclusion Criteria:

* prior incontinence surgery
* need of concomitant surgery
* post void residual urine volume < 100 ml
* urinary tract anomalies
* urinary tract infection
* more than 3 urinary tract infection within last year
* more than grade 2 urogenital prolapse
* Body mass index > 35
* Radiotherapy of the pelvic region
* active malignancy
* hemophilia
* anticoagulant treatment
* neurological disorder or other disease which affects bladder function
* anticholinergic treatment
* use of duloxetine
* do not understand the purpose of the trial
* immobility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2004-04; Study Completion 2010-12

PRIMARY OUTCOMES:
Complications
Objective cure rate by stress test and pad weighing test

SECONDARY OUTCOMES:
Quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Carl G Nilsson, MD,PhD, Principal Investigator — Helsinki University, Dept Obstet Gynecol, Helsinki University Central Hospital; Carl G Nilsson, MD,PhD, Principal Investigator — University of Helsinki
Locations (1):
- Helsinki University, Dept Obstet Gynecol, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Kuuva N, Nilsson CG. A nationwide analysis of complications associated with the tension-free vaginal tape (TVT) procedure. Acta Obstet Gynecol Scand. 2002 Jan;81(1):72-7. doi: 10.1034/j.1600-0412.2002.810113.x. PMID 11942891
- [Derived] Laurikainen E, Valpas A, Aukee P, Kivela A, Rinne K, Takala T, Nilsson CG. Five-year results of a randomized trial comparing retropubic and transobturator midurethral slings for stress incontinence. Eur Urol. 2014 Jun;65(6):1109-14. doi: 10.1016/j.eururo.2014.01.031. Epub 2014 Jan 31. PMID 24508070
- [Derived] Laurikainen E, Valpas A, Kivela A, Kalliola T, Rinne K, Takala T, Nilsson CG. Retropubic compared with transobturator tape placement in treatment of urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):4-11. doi: 10.1097/01.AOG.0000249607.82768.a1. PMID 17197581
- See also: International urogynecological association — http://www.iuga.org/